CLINICAL TRIAL: NCT00592046
Title: A Phase I Trial of ZIO-101 in Hematologic Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGL1001
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Acute Leukemia; Chronic Myeloproliferative Disease; Chronic Lymphoproliferative Disease; Multiple Myeloma; Lymphoma; Poor-risk Myelodysplasia (MDS)
Keywords: Phase I; Hematologic Cancers; Blood Cancers; Leukemia; multiple myeloma; myelodysplasia (MDS); Relapsed/refractory leukemia or lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Multiple Myeloma; Lymphoma; Hematologic Neoplasms; Leukemia; Anemia, Refractory, with Excess of Blasts; Recurrence | interventions — darinaparsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: ZIO-101 (Darinaparsin)

INTERVENTIONS:
Drug: ZIO-101 (Darinaparsin) — ZIO-101 (Darinaparsin) given for five consecutive days to be repeated every 28 days for up to six months. This is a dose escalation study.
  Other Names: ZIO-101

SUMMARY:
This study uses a new investigational (not yet approved by the FDA for widespread use) drug called ZIO-101, an organic arsenical. You must be diagnosed to have relapsed/refractory leukemia or lymphoma (blood cancer) and have tried other standard therapies.

This study is designed to determine whether ZIO-101 may be given safely. The study will also test whether ZIO-101 helps to treat blood cancer.

We anticipate that approximately 22 to 35 patients will take part in this study.

Arsenic has been used as a medicinal agent for centuries in many different cultures. Most recently in the United States, an inorganic arsenic compound was approved by the FDA for the treatment of patients with relapsed acute promyelocytic leukemia (APL). However, use of inorganic arsenic is limited by a narrow range of activity and systemic toxicity, most notably of the cardiac system.

ZIO-101 is an organic arsenic derivative. In vitro testing in both the National Cancer Institute (NCI) cancer cell panel and in vivo testing in a leukemia animal model demonstrated substantial activity of SGLU against hematologic cancers. In vitro testing of SGLU using the NCI human cancer cell panel also detected activity against lung, colon and brain cancers, melanoma, and ovary and kidney cancers. Moderate activity was seen against breast and prostate cancers cells. Data suggest that organic arsenic generates reactive oxygen species in the cells to induce apoptosis and cell cycle arrest.

DETAILED DESCRIPTION:
The purpose of this study is to find answers to the following questions:

1. What is the largest dose of ZIO-101 that can be given once a day for 5 days every 4 weeks (a "cycle")?
2. What are the side effects of ZIO-101 when administered in this way?
3. After getting the drug how much of the ZIO-101 remains in the blood stream up to 8 days after the first injection?
4. Is ZIO-101 useful in reducing my blood cancer?

A series of tests will be taken throughout the study: medical history will be recorded, a physical exam performed, an electrocardiogram (EKG) (a measurement of your heart activity), blood tests. The amount of blood taken for these lab tests will equal about 2 1/2 tablespoons. In addition, a urine pregnancy test (if applicable), and a urine sample taken to test if your kidneys are working correctly. To see the current condition of your blood cancer, additional tests may need to be performed if they have not already been done recently. These tests may include: a bone marrow biopsy, special testing of your blood, a CT scan and a bone scan.

Immediately before being treated with ZIO-101, you will have another physical examination, you will also be asked about any medicines you are taking and how you are feeling. The blood tests may need to be repeated along with the EKG and the urine test. In addition, a small blood sample must be taken immediately before the injection of ZIO-101.

The injections of ZIO-101 will take approximately one hour. Following the first injection only, you will have 6 samples of blood taken at 0.5, 1, 2, 4, 8 and 12 hours. Additional blood samples will be taken prior to each dose of ZIO-101 only. You will also have repeat EKG within one hour after completing the injection. This process will be repeated for 5 consecutive days.

Your next visit will be Week 2 and at the onset of this visit, a blood sample will be taken and you will be asked how you feel. At Weeks 3 and 4, another blood sample will be taken and you will be asked how you feel.

At the end of Week 4, a new cycle begins. Immediately before being treated with ZIO-101, you will have a physical examination, you will be asked about any medicines you are taking and how you are feeling. The blood tests will be repeated along with the EKG and the urine test. In addition, any test used to measure your blood cancer will be repeated toward the end of the cycle.

You may receive up to six of these cycles.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have relapsed/refractory leukemia or lymphoma for which no standard therapies are anticipated to result in a durable remission. Relapsed/refractory leukemia/lymphoma includes acute leukemia, chronic myeloproliferative disease, chronic lymphoproliferative disease, multiple myeloma, and any type of lymphoma. Subjects with poor-risk myelodysplasia (MDS) are also candidates for this protocol. Poor risk MDS includes refractory anemia with excess blasts or excess blasts in transformation, and chronic myelomonocytic leukemia.
* ECOG performance status of ≤ 2.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial. Nursing subjects are excluded. Sexually active men must also use acceptable contraceptive methods. Pregnant and nursing subjects are excluded because the effects of ZIO-101 on a fetus or nursing child are unknown.
* Must be able and willing to give written informed consent.
* Absent rapidly progressing disease, the interval from cancer therapy should be ≥ 3 weeks. Subjects receiving hydroxyurea should be on stable dose ≥ 7 days before beginning treatment protocol. Persisting chronic toxicities from prior therapy must be ≤ grade 1.
* Subjects must have the following clinical laboratory values:

  * Serum creatinine ≤ 2 x the upper limit of normal
  * Total bilirubin ≤ 2 x the upper limit of normal.
  * Alanine aminotransferase (ALT), or aspartate aminotransferase (AST) ≤ 3 x the upper limit of normal.
* QTc interval < 450-470 mSec

Exclusion Criteria:

Subjects with any one of the following criteria will not be eligible for study participation:

* Patients with indolent and stable myeloma, MDS or CLL not requiring therapy are not eligible.
* Central nervous system (CNS) involvement with cancer.
* Uncontrolled active infection of any kind. Subjects with infections that are under active treatment with antibiotics and whose infections are controlled may be entered to the study.
* Active heart disease including myocardial infarction within previous 6 months; symptomatic coronary artery disease; any type of chronic, ongoing arrhythmias; or uncontrolled congestive heart failure.
* Concomitant therapy for hematologic cancer (except hydroxyurea).
* NYHA functional class ≥ 3, myocardial infarction ≤ 6 mo or uncontrolled cardiac arrhythmia other than asymptomatic atrial fibrillation; QTc ≥450msec; AV-block ≥ grade-2 or Left Bundle Branch Block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Response Rate | 6 months

SECONDARY OUTCOMES:
The RECIST criteria will be used for patients with all leukemias and myelodysplastic syndromes. | 6 months
Patients with lymphoma or myeloma will be assessed by the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas. | 6 months
EBMT, IBMTR and ABMTR criteria for definition of response, relapse and progression in patients with multiple myeloma . | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Houston, Texas, United States